CLINICAL TRIAL: NCT05347641
Title: A Single-arm, Prospective, Single-center, Phase II Clinical Study of Penpulimab Combined With RMA in the Treatment of Newly Diagnosed Primary CNS Lymphoma
Brief Title: Penpulimab Combined With RMA Treatment of Primary Diagnosis of Primary Central Nervous System Lymphoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-GL1-AF03
Record Dates: First submitted 2022-04-20; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Primary Central Nervous System Lymphoma
MeSH Terms: interventions — penpulimab; Rituximab; Methotrexate; Cytarabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Penpulimab combined with RMA was used for first-line treatment of PCNSL (Experimental): One course of treatment was performed every 21 days. After 3 courses, patients underwent cranial MR+ whole-body enhanced CT for disease assessment. Patients who did not achieve partial response (PR) were withdrawn, and patients who achieved PR or complete response (CR)/uncertain CR (CRu) were given 3 courses of treatment.
  Interventions: Drug: Penpulimab

INTERVENTIONS:
Drug: Penpulimab — Penpulimab + RMA regimen:
  Rituximab 375 mg/m2 d0 iv Methotrexate (MTX) 3.5g/m2 drip D1 Cytarabine * (ARA-C) 1-2g/m2 q12H D2-3 iv Penpulimab 200 mg iv D5
  Other Names: rituximab; Methotrexate; Cytarabine

SUMMARY:
To explore PFS, ORR (CR/CRu+PR), OS and side effects of piamprizumab combined with RMA in newly diagnosed PCNSL, so as to clarify the value of piamprizumab combined with RMA in the first-line treatment of PCNSL patients, and to clarify the clinical and biological factors affecting the efficacy

ELIGIBILITY:
Inclusion Criteria:

* For initial PCNSL confirmed by pathological tissue, the diagnostic criteria were based on WHO diagnostic criteria in 2016
* Head MR (plain scan + enhancement) performed 28 days prior to study enrollment should show the presence of at least one measurable lesion in two vertical directions (according to 2014 Lugano criteria); Or abnormal cerebrospinal fluid examination (including cerebrospinal fluid protein, cells, NGS), or ophthalmologic examination confirmed the retina, vitreous lesions
* PS score was 0~4 according to ECOG

Exclusion Criteria:

* Organs or lymph nodes outside the central nervous system are involved
* Patients with a second primary tumor (other than non-melanoma skin cancer in situ, superficial bladder cancer, cervical cancer in situ, gastrointestinal intramucosal cancer or breast cancer that has been cured and has not recurred within 5 years)
* Has a history of allergic disease, severe drug allergy, or is known to be allergic to any component of a macromolecular protein preparation or penpulimab injection prescription
* Prior treatment with anti-PD-1 antibody, anti-PD-L1 antibody, anti-PD-L2 antibody, anti-CTLA-4 antibody, or CAR T cell therapy (or any other antibody that acts on T cell co-stimulation or checkpoint pathways)
* A severe acute or chronic infection requiring systemic treatment
* The investigator believes that the subjects may have other factors that affect the efficacy or safety evaluation of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
2-year PFS rate of PCNSL patients treated with penpulimab combined with RMA | 2 years

SECONDARY OUTCOMES:
ORR, 2-year OS rate and safety of penpurlimab combined with RMA in first-line treatment of PCNSL patients | 2 years

IPD SHARING:
Plan to Share IPD: No